CLINICAL TRIAL: NCT05641038
Title: Comparison Of The Efficiencies Of Peloid Therapy and Paraffine Treatments In Patients With Hallux Rigidus
Brief Title: Comparison Of The Efficiencies Of Peloid and Paraffine Treatments In Patients With Hallux Rigidus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Seda ÇIRA, Principal Investigator, Doctor, Konya Meram State Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: beyhekimtrh
Record Dates: First submitted 2022-01-02; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Hallux Rigidus
Keywords: hallux rigidus; paraffin therapy; peloid therapy; exercise
MeSH Terms: conditions — Hallux Rigidus; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study was designed as prospective, case-control and hospital-based.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Peloid treatment (Active Comparator): The patients in the first group; Peloid was applied to both feet at 42 °C for 2 weeks, 5 days a week, 10 sessions in total, 20 minutes each session.
  Interventions: Other: Peloid treatment
- Group 2 Paraffin treatment (Active Comparator): The patients in the second group were given paraffin treatment on both feet by dipping method, for 2 weeks, 5 days a week, 10 sessions in total, 20 minutes each session.
  Interventions: Other: Paraffin treatment

INTERVENTIONS:
Other: Peloid treatment — The patients in the first group; Peloid was applied to both feet at 42 °C for 2 weeks, 5 days a week, 10 sessions in total, 20 minutes each session. Peloid was applied in a layer of approximately 1.5-2 cm thick, then the foot was wrapped in a nylon bag and covered with a towel. After 20 minutes of application, the peloid layer was removed and disposed of in medical waste. The treatment area was cleaned with soft cloths moistened with hot water and the session was ended. In addition to peloid therapy, a home exercise program including joint range of motion, stretching and strengthening exercises for the 1st MTF with 3 sets of 10 repetitions was described for the patients to do simultaneously.
  Arms: Group 1 Peloid treatment
Other: Paraffin treatment — The patients in the second group were given paraffin treatment on both feet by dipping method, for 2 weeks, 5 days a week, 10 sessions in total, 20 minutes each session. After the foot was dipped and removed 10 times, it was wrapped in a nylon bag and left for 20 minutes. Then the paraffin was peeled off the feet and disposed of in medical waste. Likewise, a home exercise program including joint range of motion, stretching and strengthening exercises for the 1st MTF with 3 sets of 10 repetitions was described for them to do simultaneously.
  Arms: Group 2 Paraffin treatment

SUMMARY:
In the study, the effects of peloid and paraffin treatments applied to symptomatic hallux rigidus patients on pain, functional status, quality of life and joint range of motion were evaluated and their effectiveness was compared.

DETAILED DESCRIPTION:
Hallux rigidus(HR); It is a pathology seen in the first Metatarsophalangeal (MTF) joint, characterized by pain, dorsal osteophytes, and dorsiflexion difficulties due to progressive degenerative arthritis. (1) The most common deformity of the first MTF joint is hallux valgus, and the second most common deformity is HR. Its incidence is higher in women than in men.(2, 3) Clinically, HR typically has insidious onset pain in the MTF joint when walking and a decrease in joint range of motion (ROM).(4) X-rays are used in radiological evaluation; narrowing of the joint space, osteophytes in the head of the metatarsal and proximal phalanx, and deterioration of the nonuniform cartilage can be observed. (5) The Coughlin and Shurnas staging system, which was created in 1999 by adding range of motion and patient's symptoms to radiological findings, is one of the most preferred.(6) This staging system was used in the staging of the patients in our study.

Treatment of HR varies according to the patient's clinic and the stage of the disease. The preferred treatment option in the early period is conservative methods. Nonsteroidal anti-inflammatory drugs (NSAI) can be used to alleviate synovitis and joint inflammation. (7) Other non-operative treatment modalities of HR include physical therapy modalities (hot-cold therapy, electrotherapy), exercise (stretching-strengthening exercises), bracing, manipulation. ..etc.(8,9) However, hard-soled shoes with a deep and wide front are recommended for activity modification and reduction of dorsal compression. Dynamic splinting can be applied to patients to increase dorsiflexion. (10) Intra-articular steroid, hyaluronic acid or platelet rich plasma (PRP) injection can be applied to patients who do not respond to these treatments. (8,11) There are many surgical methods defined for the treatment of HR. These; joint debridement, osteophyte excision, resection arthroplasty, interposition arthroplasty, cheilectomy, proximal phalangeal or metatarsal osteotomy, arthrodesis and implant arthroplasty.(12) Paraffin therapy is one of the superficial heating treatment methods. The melting point of solid paraffin is 70-80 degree. This temperature is reduced to 50-55 degree by adding 1/4 - 1/7 liquid paraffin or mineral oil. (13) There are two application methods, immersion and brushing. The immersion method is applied to the extremities, that is, for the hands, feet and arms. Brushing method is more suitable for other parts of the body such as hips, shoulders and back. With paraffin treatment, a very intense heat transfer is provided to the body. It is known that paraffin therapy also creates an increase in temperature in the joint capsule and muscles. (14) Peloids are mixtures of organic and/or inorganic substances formed as a result of biological, climatological and/or geological events. Peloid therapy is a special balneotherapy method made with natural mud.(15,16) Peloids can be applied in the form of baths (full, half, sitting and extremity baths), packs, tampons, kneading and masks. The most commonly used method in peloid therapy is packaged applications. (17) They provide relief of muscle spasm and reduction of pain with their mechanical effects. In the venous system, blood is directed towards the heart from the peripheral veins. There is a decrease in peripheral vein tone, a decrease in diastolic pressure, and a slight increase in systolic blood pressure. Vasodilation occurs in the relevant deep parts of the body with the cutaneous reflex that arises with stimulation in the parts of the body that come into contact with the peloid, muscle spasm, which is mostly thought to be due to ischemia, is resolved by thermic effect and vasodilation, vasodilation helps to clear the metabolic wastes that may cause pain from the tissue and as a result, the pain disappears. It causes relaxation in muscles, soft tissues (such as tendons, ligaments, fascia and joint capsule), raises the pain threshold at nerve endings and provokes a series of neuroendocrine reactions. In addition, hot applications have an anti-inflammatory effect in chronic inflammations. (16,18) The organic (bitumen, pectin, cellulose, lignin, humin, sulfoglycolipids, humic, fulvic and ulmic acids) and inorganic (sulphur, sodium and magnesium chloride, sulfate, iodine, bromine, zinc and selenium) substances contained in the peloid also cause many effects in the body. . The absorption of these substances through the skin causes vasodilation, relaxation in smooth muscles, inhibition of inflammation in Langerhans cells in the skin, stopping the breakdown of arachidonic acid into prostaglandins, suppressing hyaluronidase activity, and antioxidant, antiviral and anti-inflammatory effects.(19,20) Thermal mud baths activate the pathway. It has been shown to cause an increase in various hormones, a decrease in important mediators in inflammation and pain, a decrease in mediators involved in cartilage destruction, and an increase in antioxidant activity.(21) It is used in the treatment of many diseases; especially such as chronic low back and neck pain, degenerative joint diseases, soft tissue rheumatism, discopathies and arthralgias. (22-25) There are no comprehensive and adequate studies conducted in patients with symptomatic HR with paraffin administration and peloid therapy. It is thought that peloid and paraffin treatments may have a positive effect on pain, functional status and quality of life in patients with HR. The aim of this study; to investigate the effectiveness of peloid and paraffin treatments on pain, functional status and quality of life in the treatment of symptomatic HR and to compare the results.

In the study, patients who applied to our Health Sciences University Konya Physical Medicine and Rehabilitation polyclinics and were diagnosed with HR clinically and/or radiologically and sent for treatment were examined. Among these patients, 80 patients were included in the study according to the inclusion and exclusion criteria. The patients were divided into two groups of 40 each as peloid therapy and paraffin therapy. Detailed histories of the patients were taken and their sociodemographic and clinical characteristics were recorded. Peloid treatment was given to the first group for 2 weeks, 5 days a week, for a total of 10 sessions. The second group was given paraffin treatment for 2 weeks, 5 days a week, for a total of 10 sessions. A home exercise program including ROM, stretching and strengthening exercises was added to both treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Pain-limitation in the 1st MTF joint for three months or longer,
* Being over 35 years old,
* 3 or more severe pain according to VAS,
* Localized tenderness over the 1st MTF on palpation.

Exclusion Criteria:

* Having neuropathic or radicular pain,
* History of acute trauma,
* Previous surgical intervention on the foot or non-operative treatment within 6 months (corticosteroid injection, physical therapy applications, shoe modifications, etc.),
* Having rheumatological diseases such as rheumatoid arthritis, psoriatic arthritis, gout,
* Having a malignancy,
* Having a progressive neurological disease that causes sensory defects,
* Being allergic to peloid therapy,
* Being pregnant
* Having a communication problem.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Descriptive Characteristics of the Patients | Just before the treatment, both groups will be asked in the form of a short questionnaire.
  A short questionnaire was created to determine the sociodemographic characteristics of the patients.
Evaluation of Pain Severity | Patients were evaluated just before treatment. (1st measurement)
  The pain level of the patients was determined by a visual analog scale(VAS). The patient was asked to mark the value corresponding to resting pain and pain during walking on the scale.
Evaluation of Functionality and Quality of Life | Patients were evaluated just before treatment. (1st measurement)
  Foot-ankle outcome score (FAOS) is an international questionnaire used to assess
Evaluation of Quality of Life | Patients were evaluated just before treatment. (1st measurement)
  Quality of life was evaluated with the SF-36 health questionnaire. The SF-36 is a form of 36 questions consisting of 8 subgroups, which is used to measure the general quality of life. It has eight subscales (general health, physical function, physical condition, pain, life functions, social functions, emotional status, mental health) and 2 specific scales (mental health and physical health).
Joint Range of Motion Measurement | Patients were evaluated just before treatment. (1st measurement)
  Dorsiflexion and plantarflexion angles of the 1st MTP joint in both feet of the patients were measured with a goniometer and noted. In addition, the stages of disease for the patients were determined according to the Coughlin and Shurnas staging system.
Evaluation of Pain Severity | Patients were evaluated immediately after treatment. (2nd measurement)
  The pain level of the patients was determined by a visual analog scale(VAS). The patient was asked to mark the value corresponding to resting pain and pain during walking on the scale.
Evaluation of Functionality and Quality of Life | Patients were evaluated immediately after treatment. (2nd measurement)
  Foot-ankle outcome score (FAOS) is an international questionnaire used to assess functionality and quality of life. The Turkish validity and reliability of this form were studied. This test consists of 44 questions in total. Headings include symptoms, pain, work, and daily life, sports, and recreational activities, and quality of life.
Evaluation of Quality of Life | Patients were evaluated immediately after treatment. (2nd measurement)
  Quality of life was evaluated with the SF-36 health questionnaire. The SF-36 is a form of 36 questions consisting of 8 subgroups, which is used to measure the general quality of life. It has eight subscales (general health, physical function, physical condition, pain, life functions, social functions, emotional status, mental health) and 2 specific scales (mental health and physical health).
Joint Range of Motion Measurement | Patients were evaluated immediately after treatment. (2nd measurement)
  Dorsiflexion and plantarflexion angles of the 1st MTP joint in both feet of the patients were measured with a goniometer and noted. In addition, the stages of disease for the patients were determined according to the Coughlin and Shurnas staging system.
Evaluation of Pain Severity | The patients were evaluated 1 month after the treatment. (3rd measurement)
  The pain level of the patients was determined by a visual analog scale(VAS). The patient was asked to mark the value corresponding to resting pain and pain during walking on the scale.
Evaluation of Functionality and Quality of Life | The patients were evaluated 1 month after the treatment. (3rd measurement)
  Foot-ankle outcome score (FAOS) is an international questionnaire used to assess functionality and quality of life. The Turkish validity and reliability of this form were studied. This test consists of 44 questions in total. Headings include symptoms, pain, work, and daily life, sports, and recreational activities, and quality of life.
Evaluation of Quality of Life | The patients were evaluated 1 month after the treatment. (3rd measurement)
  Quality of life was evaluated with the SF-36 health questionnaire. The SF-36 is a form of 36 questions consisting of 8 subgroups, which is used to measure the general quality of life. It has eight subscales (general health, physical function, physical condition, pain, life functions, social functions, emotional status, mental health) and 2 specific scales (mental health and physical health).
Joint Range of Motion Measurement | The patients were evaluated 1 month after the treatment. (3rd measurement)
  Dorsiflexion and plantarflexion angles of the 1st MTP joint in both feet of the patients were measured with a goniometer and noted. In addition, the stages of disease for the patients were determined according to the Coughlin and Shurnas staging system.

CONTACTS AND LOCATIONS:
Overall Officials: seda çıra, Principal Investigator — assistant doctor
Locations (1):
- Konya Beyhekim Training and Research Hospital Physical Medicine and Rehabilitation Clinic, Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wülker NJIA, Zollinger-Kies H: Fußchirurgie. Hallux rigidus. 2004;1:99-103.
- [Background] Berlet GC, Hyer CF, Lee TH, Philbin TM, Hartman JF, Wright ML. Interpositional arthroplasty of the first MTP joint using a regenerative tissue matrix for the treatment of advanced hallux rigidus. Foot Ankle Int. 2008 Jan;29(1):10-21. doi: 10.3113/FAI.2008.0010. PMID 18275731
- [Background] Thermann H, Becher C, Kilger RJTiF, Surgery A. Hallux rigidus treatment with cheilectomy, extensive plantar release, and additional microfracture technique. 2004;3(4):210-5.
- [Background] Dülgeroğlu TC, DEMİRKIRAN ND, Erduran M. İleri evre halluks rijiduslu hastalarda yerli üretim total eklem artroplastisi ile tedavi sonuçlarımız. Pamukkale Tıp Dergisi.12(2):215-24.
- [Background] Uzunca KJTJoPM, Dergisi RTFTvR. Ayak Bileği ve Ayak Osteoartritleri. 2009;55.
- [Background] Coughlin MJ, Shurnas PS. Hallux rigidus. Grading and long-term results of operative treatment. J Bone Joint Surg Am. 2003 Nov;85(11):2072-88. PMID 14630834
- [Background] Meriç G, Budeyri A, Başdelioğlu K, Demir A, UYSAL AEJBSBD. HALLUKS RİJİDUSTA KULLANILAN TEDAVİ SEÇENEKLERİ.1(2):85-9.
- [Background] Zammit GV, Menz HB, Munteanu SE, Landorf KB, Gilheany MF. Interventions for treating osteoarthritis of the big toe joint. Cochrane Database Syst Rev. 2010 Sep 8;(9):CD007809. doi: 10.1002/14651858.CD007809.pub2. PMID 20824867
- [Background] Polzer H, Polzer S, Brumann M, Mutschler W, Regauer M. Hallux rigidus: Joint preserving alternatives to arthrodesis - a review of the literature. World J Orthop. 2014 Jan 18;5(1):6-13. doi: 10.5312/wjo.v5.i1.6. eCollection 2014 Jan 18. PMID 24649409
- [Background] Kalish S, Willis FBJTF, Journal AO. Hallux limitus and dynamic splinting: a retrospective series. 2009;2(4):1.
- [Background] OKUR SÇ, FİRDİN F, ÖZTÜRK SK, EDEMCİ ŞJBTT, Regülasyon ve Nöral Terapi Dergisi. HALLUKS RİJİDUS TEDAVİSİNDE MANUAL MOBİLİZASYON TEKNİKLERİNİN ETKİNLİĞİNİN DEĞERLENDİRİLMESİ: VAKA SERİSİ.12(3):14-7.
- [Background] Kılıçoğlu Ö. Ayak başparmağının hastalıkları: Halluks valgus ve halluks rigidus.
- [Background] Stillwell G. General principles of thermotherapy. Therapeutic Heat and Cold: E. Licht New Haven (Conn.); 1965. p. 232-65.
- [Background] Oğuz h. Oğuz H, Dursun E, Dursun N, Tıbbi Rehabilitasyon. Öztürk C, Akşit R, Tedavide sıcak ve soğuk. Nobel tıp kitabevi, 2004; 333-353
- [Background] UN Ö. Kaplıca Tedavisi. In: Tuna N, Eds. Romatizmal Hastalıklar. Ankara: Hacettepe Taş Kitapçılık; 1994. s. 229-42.
- [Background] H. G. Peloidoterapi, Etki, Mekanizması ve Uygulama Yöntemleri. İçinde Karagülle M, editor. Tıbbi Ekoloji ve Hidroklimatoloji. İstanbul: Nobel Tıp Kitabevleri; 2013. 13-18. .
- [Background] M.Z. K. Kaplıca Tedavisi, Balneoterapi ve Klimaterapi. İçinde Doğan M Karagülle MZ, editör. Kaplıca Tıbbı ve Türkiye Kaplıca Rehberi. İstanbul: Nobel Tıp kitabevleri. 2002. 1-22.
- [Background] MZ K. H G. Peloidler, In: Karagülle MZ (eds). Balneoloji ve Kaplıca Tıbbı, Nobel Tıp Kitabevleri, p: 97-112, İstanbul, 2002 40.
- [Background] Odabasi E, Turan M, Erdem H, Tekbas F. Does mud pack treatment have any chemical effect? A randomized controlled clinical study. J Altern Complement Med. 2008 Jun;14(5):559-65. doi: 10.1089/acm.2008.0003. PMID 18564957
- [Background] Fraioli A, Serio A, Mennuni G, Ceccarelli F, Petraccia L, Fontana M, Grassi M, Valesini G. A study on the efficacy of treatment with mud packs and baths with Sillene mineral water (Chianciano Spa Italy) in patients suffering from knee osteoarthritis. Rheumatol Int. 2011 Oct;31(10):1333-40. doi: 10.1007/s00296-010-1475-5. PMID 20390281
- [Background] Bellometti S, Richelmi P, Tassoni T, Berte F. Production of matrix metalloproteinases and their inhibitors in osteoarthritic patients undergoing mud bath therapy. Int J Clin Pharmacol Res. 2005;25(2):77-94. PMID 16060398
- [Background] Codish S, Abu-Shakra M, Flusser D, Friger M, Sukenik S. Mud compress therapy for the hands of patients with rheumatoid arthritis. Rheumatol Int. 2005 Jan;25(1):49-54. doi: 10.1007/s00296-003-0402-4. Epub 2003 Nov 14. PMID 14618372
- [Background] Flusser D, Abu-Shakra M, Friger M, Codish S, Sukenik S. Therapy with mud compresses for knee osteoarthritis: comparison of natural mud preparations with mineral-depleted mud. J Clin Rheumatol. 2002 Aug;8(4):197-203. doi: 10.1097/00124743-200208000-00003. PMID 17041359
- [Background] Elkayam O, Ophir J, Brener S, Paran D, Wigler I, Efron D, Even-Paz Z, Politi Y, Yaron M. Immediate and delayed effects of treatment at the Dead Sea in patients with psoriatic arthritis. Rheumatol Int. 2000;19(3):77-82. doi: 10.1007/s002960050107. PMID 10776684
- [Background] Ardic F, Ozgen M, Aybek H, Rota S, Cubukcu D, Gokgoz A. Effects of balneotherapy on serum IL-1, PGE2 and LTB4 levels in fibromyalgia patients. Rheumatol Int. 2007 Mar;27(5):441-6. doi: 10.1007/s00296-006-0237-x. PMID 17033835